CLINICAL TRIAL: NCT05831085
Title: A Comparison of Imaging- and Physiology-Guided State-of-the-Art Percutaneous Coronary Intervention and Coronary-Artery Bypass Grafting in Patients With Diabetes and Three-Vessel Coronary Artery Disease: DEFINE-DM Trial (Diabetes-Centered Evaluation of Revascularization Strategy of Functional and Imaging-CombiNEd State-of-the-Art Percutaneous Coronary Intervention or Coronary-Artery Bypass Grafting in Patients With Diabetes Mellitus and Multivessel Coronary Artery Disease)
Brief Title: Diabetes-Centered Evaluation of Revascularization Strategy of Functional and Imaging-CombiNEd State-of-the-Art Percutaneous Coronary Intervention or Coronary-Artery Bypass Grafting in Patients With Diabetes Mellitus and Multivessel Coronary Artery Disease
Acronym: DEFINE-DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Cardiology, Asan Medical Center Heart Institute, Valvular Heart Disease Center, Ischemic Heart Disease Center, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMCCV2023-03
Record Dates: First submitted 2023-04-04; First posted 2023-04-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Stenosis
Keywords: Multivessel Coronary Artery Disease; state of the art; State-of-the-Art Percutaneous Coronary Intervention; Coronary-Artery Bypass Grafting; Diabetes Mellitus
MeSH Terms: conditions — Coronary Stenosis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging- and Physiology-Guided State-of-the-Art Percutaneous Coronary Intervention (Experimental)
  Interventions: Procedure: State-of-the-Art Percutaneous Coronary Intervention
- Coronary-Artery Bypass Grafting (Active Comparator)
  Interventions: Procedure: standard CABG

INTERVENTIONS:
Procedure: State-of-the-Art Percutaneous Coronary Intervention — supported by intracoronary imaging (e.g., intravascular ultrasound [IVUS] or optical coherence tomography [OCT]), intracoronary physiology (e.g., fractional flow reserve [FFR] or instantaneous wave-free ratio [iFR]), contemporary metallic DES (durable polymer everolimus-eluting stents; XIENCE family stent system, Abbott Vascular), guideline-directed optimal medical therapy [GDMT] with advanced cardiovascular (e.g., high-dose statin and advanced strategy of antiplatelet regimens) and anti-diabetic medications [e.g., a sodium-glucose cotransporter [SGLT]-2 inhibitors or Glucagon-like peptide-1 [GLP-1] agonists) in patients with type 2 diabetes and three-vessel coronary artery disease (CAD) (not involving left main)
  Arms: Imaging- and Physiology-Guided State-of-the-Art Percutaneous Coronary Intervention
Procedure: standard CABG — Coronary-Artery Bypass Grafting
  Arms: Coronary-Artery Bypass Grafting

SUMMARY:
The objective of this randomized study was to compare outcomes of imaging-and physiology-guided state-of-the-art percutaneous coronary intervention (PCI) to coronary artery bypass grafting (CABG) in patients with diabetes and three-vessel CAD (not involving left main).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be ≥20 years of age with angina and/or evidence of myocardial ischemia.
2. Patients with type 2 diabetes based on the need for treatment with insulin or oral hypoglycemic drugs or a confirmed elevated blood glucose level (fasting plasma glucose elevation on >1 occasion of ≥126 mg/dL [7.0 mmol/L] or 2-h postprandial of ≥200 mg/dL [11.1 mmol/L] during oral glucose tolerance test or random plasma glucose of ≥200 mg/dL [11.1 mmol/L] with classic symptoms of hyperglycemia or hyperglycemic crisis or HbA1C ≥6.5% [48 mmol/mol]).
3. Significant three-vessel CAD (defined as ≥ 50% diameter stenosis [DS] by visual estimation in each of the three major epicardial vessels or major side branches but not involving the left main coronary artery) and equivalently amenable to revascularization by means of either PCI or CABG as determined by the Heart Team at the trial site.
4. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Unprotected left main coronary artery disease.
2. The presence of complex coronary disease anatomy or lesion characteristics or other cardiac condition(s) which leads the participating interventional cardiologist to believe that PCI is not suitable (i.e. the subject should be managed with CABG or medical therapy alone).
3. Recent ST-elevation myocardial infarction(<5 days prior to randomization).
4. Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support.
5. Severe left ventricular dysfunction (ejection fraction <30%).
6. Requirement for other cardiac or non-cardiac surgical procedure (e.g., valve replacement, aorta surgery, or carotid revascularization). However, a maze procedure or pulmonary vein isolation is allowed.
7. Contraindication or inability to take aspirin or P2Y12 inhibitors (clopidogrel, ticagrelor, or prasugrel) for at least 6 months.
8. Prior CABG.
9. Extremely calcified or tortuous vessels precluding FFR measurement or intracoronary imaging evaluation.
10. More than one major epicardial vessel which is chronically occluded; enrollment of 1 Chronic total occlusion lesion is allowed.
11. Subjects requiring or who may require additional surgery (cardiac or noncardiac) within 1 year.
12. End-stage renal disease requiring renal replacement therapy.
13. Liver cirrhosis.
14. Pregnant and/or lactating women.
15. Concurrent medical condition with a limited life expectancy of less than 2 years.
16. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period. However, where at least one or more conditions are satisfied, it could be an exception according to an investigator's discretion;

1) Participated in the observational study expected no effect on the safety and/or effectiveness evaluation of this trial.

2) Screening failed before any interventional factor is involved.

3) Participated in academic trials like strategic comparison studies conducted under standard therapy provided that there is no additional risk or a specific procedure to a subject and no interference between this trial and other studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The event rate of major adverse cardiac or cerebrovascular events | 2 years
  Major adverse cardiac or cerebrovascular events (MACCE) were defined as a composite of hard clinical endpoints of death from any causes, myocardial infarction, or stroke.

SECONDARY OUTCOMES:
The event rate of death from any cause | 5 years
The event rate of myocardial infarction | 5 years
The event rate of repeat revascularization | 5 years
The event rate of stroke | 5 years
The event rate of composite of death from any causes, cardiovascular causes, or noncardiovascular causes | 5 years
The event rate of myocardial infarction | 5 years
  any, spontaneous or procedural
The event rate of composite of death or myocardial infarction | 5 years
The event rate of composite of death, myocardial infarction, stroke or repeat revascularization | 5 years
The event rate of stent thrombosis | 5 years
  by an Academic Research Consortium (ARC) definition
The event rate of symptomatic graft occlusion or stenosis | 5 years
The event rate of bleeding complications | 5 years
  BARC (Bleeding Academic Research Consortium) criteria
The event rate of periprocedural major adverse events | 5 years
  Periprocedural major adverse events means major arrhythmia, any unplanned surgery or therapeutic radiologic procedure, development of acute renal failure, sternal wound dehiscence, infection requiring antibiotics, prolonged intubation (>48 hours), post-pericardiotomy syndrome, etc.
Length of hospital stay | 7 days
The event rate of rehospitalization | 7 days
  any, cardiac, or noncardiac causes
The change of functional class | 1, 6, 12, 18, 24, 36, 60 months
  Assessed by The Canadian Cardiovascular Society (CCS) Angina Score Classification.
  The minimum and maximum values are 1 and 4 respectively. A higher score of CCS angina score classification means severe exertional angina.
The change of angina-related quality of life index by the Seattle Angina Questionnaire [SAQ] | 1, 12, 24, 36, 60 months
  The SAQ is a disease-specific patient-reported outcome (PRO) with 5 domains.
  The minimum and maximum values are 0 and 100 respectively. A lower score represents poor health status and a high score represents good health status.
The change of angina-related quality of life index by the EQ-5D | 1, 12, 24, 36, 60 months
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group.
  The minimum and maximum values are 5 and 15 respectively. A higher score of EQ-5D means a low quality of life.
The number of anti-anginal medications used | 1, 6, 12, 18, 24, 36, 60 months
Total healthcare costs and cost-effectiveness assessed using total medical expenditures and incremental cost-effectiveness ratio (ICER) | 1, 6, 12, 18, 24, 36, 60 months
  Total medical cost will be calculated using predefined cost components related to the index revascularization procedure (PCI or CABG) and subsequent healthcare utilization. The list of cost items includes (but is not limited to): diagnostic catheters, guide catheters, guidewires, balloons, stents, adjunctive devices (e.g., rotablation system, intravascular lithotripsy), professional procedure fees, CABG-related graft categories, hospitalization cost per day (Intensive care unit and ward), and non-invasive cardiac tests. Total costs will be aggregated for each participant and compared between study groups at each scheduled time point.
  Cost-effectiveness will be assessed using the incremental cost-effectiveness ratio (ICER), calculated as the difference in total costs divided by the difference in clinical effectiveness between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, Study Chair — Asan Medical Center
Locations (27):
- Palo Alto VA Medical Center, Palo Alto, California, United States
- China (2):
  - Fuwai Hospital, Chinese Academy of Medical Sciences (CAMS), Beijing
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou
- India (2):
  - Medanta - The Medicity, Gurugram
  - Fortis Escorts Heart Institute, New Delhi
- Sarawak Heart Centre, Kota Samarahan, Malaysia
- University Clinical Center of Serbia, Belgrade, Serbia
- National Heart Centre Singapore (NHCS), Singapore, Singapore
- South Korea (17):
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Dong-A Medical Center, Pusan
  - Asan Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
- National Taiwan University Hospital, Taipei, Taiwan
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided